CLINICAL TRIAL: NCT02651675
Title: AAV8-mediated Low Density Lipoprotein Receptor (LDLR) Gene Replacement in Subjects With Homozygous Familial Hypercholesterolemia (HoFH)
Brief Title: A Gene Therapy Study for Homozygous Familial Hypercholesterolemia (HoFH)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Terminated by Sponsor for Business Reasons
Sponsor: REGENXBIO Inc. (Industry)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: FHGT002; P01HL059407 (NIH)
Record Dates: First submitted 2016-01-04; First posted 2016-01-11 (Estimated); Results first posted 2023-07-13 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-06

CONDITIONS: Homozygous Familial Hypercholesterolemia (HoFH)
Keywords: LDL Receptors; Gene therapy; Metabolic Diseases; Rare diseases; Genetic Diseases; Atherosclerosis; cardiovascular disease
MeSH Terms: conditions — Homozygous Familial Hypercholesterolemia; Hyperlipoproteinemia Type II; Metabolic Diseases; Rare Diseases; Genetic Diseases, Inborn; Atherosclerosis; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: dose escalation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): 2.5E12 (genome copies)/kg (kilogram) body weight (E means the exponential constant)
  Interventions: Genetic: AAV directed hLDLR gene therapy
- Cohort 2 (Experimental): 7.5E12 GC/kg body weight
  Interventions: Genetic: AAV directed hLDLR gene therapy
- Cohort 2 Expansion (Experimental): 7.5E12 GC/kg body weight
  DSMB (Data Safety Monitoring Board) approved expansion of Dose 2 cohort, 3 additional subjects enrolled and received prophylactic corticosteroids
  Interventions: Genetic: AAV directed hLDLR gene therapy

INTERVENTIONS:
Genetic: AAV directed hLDLR gene therapy — AAV directed hLDLR gene therapy is a novel adeno-associated viral (AAV8) vector with human low-density lipoprotein receptor (hLDLR) gene

SUMMARY:
This first-in-human study is intended to evaluate the safety and preliminary effectiveness of AAV (Adeno-associated virus)-based liver-directed gene therapy in the treatment of adults with Homozygous Familial Hypercholesterolemia (HoFH).

DETAILED DESCRIPTION:
Homozygous Familial Hypercholesterolemia (HoFH) is a rare genetic metabolic disorder characterized by absent or severely reduced capacity to catabolize circulating LDL (Low density lipoprotein) particles by the hepatic LDL receptor. As a consequence, HoFH subjects present abnormal total plasma cholesterol (LDL-C) levels, resulting in severe atherosclerosis often leading to early onset of cardiovascular disease. Early initiation of aggressive treatment for these patients is therefore essential. Unfortunately, despite existing therapies, treated LDL-C (Low density lipoprotein cholesterol) levels could remain well above acceptable levels. Thus, the functional replacement of the defective LDLR via AAV-based liver-directed gene therapy may be a viable approach to treat this disease and improve response to current lipid-lowering treatments. This first-in-human study is intended to evaluate the safety of this gene therapy investigational product and assess preliminary evidence of efficacy using plasma LDL-C levels as a surrogate biomarker for human LDLR transgene expression.

Subjects may be asked to participate in an optional kinetics study to assess the metabolic mechanism by which LDL-C is reduced.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years of age.
* Untreated and/or treated LDL-C levels and clinical presentation consistent with the diagnosis of homozygous FH (Familial hypercholesterolemia)
* Molecularly defined LDLR mutations at both LDLR alleles.
* A baseline serum AAV8 NAb (Neutralizing antibody) titer ≤ 1:10.

Exclusion Criteria

* Unwilling to wash out of the following lipid lowering therapies for the pre-specified time period:

  1. niacin > 250 mg/day: within 6 weeks of baseline
  2. fibrates: within 4 weeks of baseline
  3. lomitapide: within 8 weeks of baseline
  4. mipomersen: within 24 weeks of baseline
* History of cirrhosis or chronic liver disease based on documented histological evaluation or non-invasive imaging or testing.
* Abnormal liver function tests (LFTs) at screening (AST (Aspartate aminotransferase) or ALT (Alanine aminotransferase) > 2 × upper limit of normal (ULN) and/or Total Bilirubin of > 1.5 × ULN

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2020-11-27 (Actual); Study Completion 2020-11-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (5):
  - Boca Raton location, Boca Raton, Florida
  - Kansas City Location, Kansas City, Kansas
  - Portland location, Portland, Oregon
  - Philadelphia Location, Philadelphia, Pennsylvania
  - Nashville location, Nashville, Tennessee
- Montreal location, Montreal, Quebec, Canada
- Italy (2):
  - Palermo location, Palermo, PA
  - Rome location, Roma, RM
- Rotterdam location, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: 2.5E12 GC (genome copies)/kg (kilogram body weight (E means exponential constant)
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 2 Expansion
Started | 3 | 3 | 3
Completed | 3 | 3 | 2
Not Completed | 0 | 0 | 1
Not completed — Death | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1: 2.5E12 GC/kg body weight
  Single intravenous (IV) dose of human Low Density Lipoprotein Receptor (LDLR) Gene Therapy
  AAV directed hLDLR gene therapy: a novel adeno-associated viral (AAV8) vector with human low-density lipoprotein receptor (hLDLR) gene
- Cohort 2: 7.5E12 GC/kg body weight
  Single intravenous (IV) dose of human Low Density Lipoprotein Receptor (LDLR) Gene Therapy
  AAV directed hLDLR gene therapy: a novel adeno-associated viral (AAV8) vector with human low-density lipoprotein receptor (hLDLR) gene
- Cohort 2 Expansion: 7.5E12 GC/kg body weight
  DSMB (Data Safety Monitoring Board) approved expansion of Dose 2 cohort, 3 additional subjects enrolled and received prophylactic corticosteroids
  Single intravenous (IV) dose of human Low Density Lipoprotein Receptor (LDLR) Gene Therapy
  AAV directed hLDLR gene therapy: a novel adeno-associated viral (AAV8) vector with human low-density lipoprotein receptor (hLDLR) gene
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 2 Expansion | Total
Number analyzed (Participants) | 3 | 3 | 3 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 3 | 9
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 3
  Male | 2 | 2 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 2 | 3 | 3 | 8
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 1 | 3 | 3 | 7
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 0 | 1 | 0 | 1
  Netherlands | 0 | 0 | 2 | 2
  United States | 3 | 2 | 0 | 5
  Italy | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With IP (Investigational Product) Related Adverse Events
Description: Physical examinations; Clinical laboratory parameters; and adverse event reporting
Time Frame: Up to 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 2 Expansion
Number analyzed (Participants) | 3 | 3 | 3
Participants | 1 | 3 | 2

2. Secondary Outcome: Percent Change in LDL-C
Description: Percent change in LDL-C compared to baseline
Time Frame: 18 weeks, 12 weeks for cohort 1 only, compared to baseline
Measure: Mean (Standard Deviation); unit: percentage of change from baseline
Arm/Group | Cohort 1 | Cohort 2 | Cohort 2 Expansion
Number analyzed (Participants) | 3 | 3 | 3
percentage of change from baseline | 7.21 (12.24) | 27.35 (32.51) | 8.98 (31.34)

3. Secondary Outcome: Percent Change in Lipid Parameters Compared to Baseline Values
Description: total cholesterol (TC); non-high density lipoprotein cholesterol (non-HDL-C); HDL-C; fasting triglycerides (TG); overflow density lipoprotein cholesterol (VLDL-C); lipoprotein(a) (Lp(a)); apolipoprotein B (apoB) and apolipoprotein A-I (apo A-I)
Time Frame: 18 weeks, 12 weeks for cohort 1 only, compared to baseline
Measure: Mean (Standard Deviation); unit: percentage of change from baseline
Arm/Group | Cohort 1 | Cohort 2 | Cohort 2 Expansion
Number analyzed (Participants) | 3 | 3 | 3
percentage of change from baseline
  apolipoprotein B (apoB) | 4.53 (9.61) | 21.15 (25.21) | 11.36 (26.43)
  total cholesterol (TC) | 7.89 (15.72) | 24.91 (34.45) | 7.17 (37.35)
  overflow density lipoprotein cholesterol (VLDL-C) | 32.63 (85.34) | 54.17 (135.53) | -5.46 (111.43)
  fasting triglycerides (TG) | 7.92 (26.43) | -9.16 (8.23) | 15.60 (10.46)
  HDL-C | 9.10 (22.58) | 7.92 (21.68) | -10.07 (25.12)
  non-high density lipoprotein cholesterol (non-HDL-C) | 8.43 (15.93) | 27.06 (36.63) | 8.26 (38.16)
  lipoprotein(a) (Lp(a)) | -0.3 (26.31) | -31.4 (16.08) | 30.3 (17.83)
  apolipoprotein A-I (apo A-I) | -2.71 (15.18) | 12.25 (18.90) | -16.18 (11.04)

4. Secondary Outcome: Number of Participants With IP Related Adverse Events
Description: Physical examinations; Clinical laboratory parameters; and adverse event reporting
Time Frame: up to 104 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 2 Expansion
Number analyzed (Participants) | 3 | 3 | 3
Participants | 1 | 3 | 2

5. Secondary Outcome: Amount of Vector Shedding, Urine
Description: Amount of virus secreted in urine
Time Frame: up to 104 weeks
Measure: Mean (Standard Deviation); unit: GC/12 μL (microliter) specimen) (urine)
Arm/Group | Cohort 1 | Cohort 2 | Cohort 2 Expansion
Number analyzed (Participants) | 3 | 1 | 1
GC/12 μL (microliter) specimen) (urine) | 25.0 (0.0) | 25.0 (NA) — No Standard Deviation could be calculated as there is only one patient assessable at this timepoint | 0 (NA) — No Standard Deviation could be calculated as there is only one patient assessable at this timepoint

6. Secondary Outcome: Amount of Vector Shedding, Plasma
Description: Amount of virus secreted in plasma
Time Frame: up to 104 weeks
Measure: Mean (Standard Deviation); unit: GC/ μg (microgram) DNA
Arm/Group | Cohort 1 | Cohort 2 | Cohort 2 Expansion
Number analyzed (Participants) | 3 | 1 | 1
GC/ μg (microgram) DNA | 50.0 (0.0) | 50.0 (NA) — No Standard Deviation could be calculated as there is only one patient assessable at this timepoint | 0.0 (NA) — No Standard Deviation could be calculated as there is only one patient assessable at this timepoint

ADVERSE EVENTS:
Time Frame: up to 104 weeks
Description: regular investigator assessment
Groups:
- Cohort 1: 2.5E12 GC/kg body weight
  Single intravenous (IV) dose of human Low Density Lipoprotein Receptor (LDLR) Gene Therapy
  AAV directed hLDLR gene therapy: A novel adeno-associated viral (AAV) vector with human low-density lipoprotein receptor (hLDLR) gene
- Cohort 2: 7.5E12 GC/kg body weight
  Single intravenous (IV) dose of human Low Density Lipoprotein Receptor (LDLR) Gene Therapy
  AAV directed hLDLR gene therapy: A novel adeno-associated viral (AAV) vector with human low-density lipoprotein receptor (hLDLR) gene
- Cohort 2 Expansion: 7.5E12 GC/kg body weight
  DSMB (Data Safety Monitoring Board) approved expansion of Dose 2 cohort, 3 additional subjects enrolled and received prophylactic corticosteroids
  Single intravenous (IV) dose of human Low Density Lipoprotein Receptor (LDLR) Gene Therapy
  AAV directed hLDLR gene therapy: A novel adeno-associated viral (AAV) vector with human low-density lipoprotein receptor (hLDLR) gene
Arm/Group | Cohort 1 | Cohort 2 | Cohort 2 Expansion
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 1/3
Serious Adverse Events (participants affected / at risk) | 2/3 | 1/3 | 1/3
Other Adverse Events (participants affected / at risk) | 2/3 | 3/3 | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=3) | Cohort 2 (N=3) | Cohort 2 Expansion (N=3)
device failure (Product Issues) | 0 (0) | 0 (0) | 1 (1) — acute failure of prosthetic aortic valve
cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
pnuemonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) — acute lung failure
acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) — shortness of breath
hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) — worsening of angina
chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) — chest pain unknown etiology
appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
hepatic enzyme increased (Investigations) | 0 (0) | 1 (1) | 0 (0) — elevated liver enzymes
Acute left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) — acute on chronic diastolic heart failure
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=3) | Cohort 2 (N=3) | Cohort 2 Expansion (N=3)
Angina Pectoris (Cardiac disorders) | 2 (4) | 0 (0) | 0 (0)
Acute Coronary Syndrome (Cardiac disorders) | 1 (2) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1)
Chest Pain (General disorders) | 1 (1) | 0 (0) | 2 (2)
Fatigue (General disorders) | 0 (0) | 1 (1) | 2 (2)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 0 (0)
Swelling Face (General disorders) | 0 (0) | 1 (1) | 1 (1)
Hepatic Enzyme Increased (Investigations) | 1 (1) | 3 (12) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to early termination of the program for business reasons, planned efficacy analysis was not possible.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-12-14): https://cdn.clinicaltrials.gov/large-docs/75/NCT02651675/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-14): https://cdn.clinicaltrials.gov/large-docs/75/NCT02651675/SAP_001.pdf